CLINICAL TRIAL: NCT01479413
Title: Mitochondria and Schizophrenia: Effects of Antipsychotic Drugs
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Tiao-Lai Huang, Head of Department of Psychiatry, Chang Gung Memorial Hospital
Other Study IDs: CMRPG891561
Record Dates: First submitted 2011-07-10; First posted 2011-11-24 (Estimated); Last update posted 2013-09-11 (Estimated); Status verified 2013-09

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Oxidative stress; Mitochondria
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Schizophrenia

SUMMARY:
The investigators will investigate

1. the relationships between oxidative stress-, apoptosis-related markers, mitochondria DNA copy numbers and the clinical psychopathology of schizophrenia, including severity of positive and negative symptoms, obesity and metabolic syndrome.
2. the relationships between aberrant mitochondria genes (single nucleotide polymorphism of D-loop region-related genes and haplogroup N9a), DISC1 gene polymorphism, and clinical phenotypes in Taiwanese populations.
3. whether these biological markers could be as clinical markers in schizophrenia for a long-term follow-up study.

DETAILED DESCRIPTION:
In past study, we had shown that there were significant differences in serum Lpo (lipid peroxidation) and Thiol levels between patients with schizophrenia and healthy controls. For patients taking risperidone, there were significant decreases in serum Thiol levels. In addition, there were also significant differences in age of onset of PPAR gamma coactivator 1α (PGC-1α) polymorphism for schizophrenia patients. Therefore, we want to know the relationships between oxidative stress-, apoptosis-related markers, mitochondria DNA copy numbers and the clinical psychopathology of schizophrenia, including severity of positive and negative symptoms, obesity and metabolic syndrome.

In past study, we also found that there were significant differences in 10 SNPs located in the D-loop region-related genes between patients and healthy controls. Three SNPs could be found in Mitomap data, but another seven SNPs not been found in the Mitomap and they could be more confirmed. In addition, Tanaka et al. found that haplogroup N9a was related to diabetes and metabolic syndrome in Asia. Therefore, we were interested to clarify the relationships between above related mitochondria genes and clinical phenotypes in Taiwanese populations,.

In addition, we also want to see whether these biological markers could be as clinical markers in schizophrenia for a long-term follow-up study.

ELIGIBILITY:
Inclusion Criteria:

1. Schizophrenic patients will be recruited in psychiatric inpatients and outpatients departments according to DSM-IV criteria by a semi-structured interview. The assessment will be done by two senior psychiatrists. The intra- rater and inter-rater reliability will be done before this project started.
2. The patients had the ability to complete the written inform consent.

Exclusion Criteria:

1. Alcohol abuse or dependence
2. Smoking more than 1 pack per day
3. Concurrent use of mood stabilizer or beta-blocker

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will be conducted in our clinical setting. By a semi-structured interview for DSM-IV criteria, about 300 schizophrenic patients will be recruited in this study.
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2009-08; Primary Completion 2012-07 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Serum oxidative stress | 15 months
  serum malondialdehyde (MDA) content, serum free thiols, serum glutathione, catalase, Superoxide dismutase, glutathione peroxidase, proapoptotic markers (bad and bax) and antiapoptotic markers (bcl-2 and bcl-x1), quantification of mitochondrial DNA
DISC1 gene polymorphism | 15 months

SECONDARY OUTCOMES:
PANSS score | 15 months
  Positive and Negative Syndrome Scale to reflect the severity of psychopathology
Obesity | 15 months
  obesity defined by body mass index (BMI)>=26.4
Metabolic syndrome | 15 months
Drug response | 15 months

CONTACTS AND LOCATIONS:
Overall Officials: Tiao-Lai Huang, M.D., Principal Investigator — Chang-Gung Memorial Hospital, Kaohsiung
Locations (1):
- Department of Psychiatry, Chang Gung Memorial Hospital, Kaohsiung City, Taiwan